CLINICAL TRIAL: NCT01167712
Title: GOG-0262: A Phase III Trial of Every-3-Weeks Paclitaxel Versus Dose Dense Weekly Paclitaxel in Combination With Carboplatin With or Without Concurrent and Consolidation Bevacizumab (NSC #704865) in the Treatment of Primary Stage II, III or IV Epithelial Ovarian, Peritoneal or Fallopian Tube Cancer and ACRIN 6695: Perfusion CT Imaging to Evaluate Treatment Response in Patients Participating in GOG-0262
Brief Title: Paclitaxel and Carboplatin With or Without Bevacizumab in Treating Patients With Stage II, Stage III, or Stage IV Ovarian Epithelial Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03812; NCI-2011-03812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0262/ACRIN 6695; 11-00374; CDR0000681448; ACRIN 6695; GOG-0262 (Other: NRG Oncology); GOG-0262 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-07

CONDITIONS: Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinofibroma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIA Ovarian Cancer AJCC V6 and v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Ovarian Cancer AJCC v6 and v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Ovarian Cancer AJCC v6 and v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (adjuvant chemotherapy suboptimally debulked) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Paclitaxel; Procedure: Therapeutic Conventional Surgery
- Arm II (neoadjuvant chemotherapy) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses. Patients undergo interval cytoreductive surgery between courses 3 and 4.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Paclitaxel; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Correlative studies
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase III clinical trial studies two different dose schedules of paclitaxel to see how well they work in combination with carboplatin with or without bevacizumab in treating patients with stage II, III or IV ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab is a type of drug called a monoclonal antibody and blocks tumor growth by stopping the growth of blood vessels that tumors need to grow. It is not yet known whether giving paclitaxel with combination chemotherapy once every three weeks is more effective than giving paclitaxel once a week in treating patients with ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the weekly paclitaxel regimen increases the time until first progression or death (progression-free survival [PFS]) compared to the every-3-week paclitaxel regimen in women with primary stage II, III or IV epithelial ovarian, peritoneal or fallopian tube cancer who are receiving carboplatin with or without bevacizumab.

SECONDARY OBJECTIVES:

I. To determine if the weekly paclitaxel increases the duration of overall survival compared to the every-3-week paclitaxel when combined with carboplatin with or without bevacizumab.

II. To compare the weekly paclitaxel to the every-3-week paclitaxel with respect to the incidence of severe or serious adverse events when it is combined with carboplatin with or without bevacizumab.

III. To compare the weekly paclitaxel to the every-3-week paclitaxel with respect to patients' self-reported quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy-Ovarian (FACT-O)-Trial Outcome Index (TOI), when paclitaxel is combined with carboplatin with or without bevacizumab. (As of 02/08/2012, the QOL portion of this study is complete; patients enrolled after this date will not have QOL assessments)

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To evaluate single nucleotide polymorphisms (SNPs) associated with progression-free survival and toxicity in advanced stage epithelial ovarian, peritoneal and fallopian tube cancer using genome wide association studies (GWAS).* II. To evaluate genomic signatures in tumor tissues which are predictive for patient survival in advanced stage epithelial ovarian, peritoneal and fallopian tube cancer.* III. To evaluate the association between serum and plasma biomarkers and response to anti-angiogenesis therapy in advanced stage epithelial ovarian, peritoneal, and fallopian tube cancer.*

NOTE: *As of 02/08/2012, the translational research (TR) portion of this study is complete; patients enrolled after this date will not have TR specimens collected.

IMAGING PRIMARY OBJECTIVES:

I. To determine whether larger changes in the tumor perfusion parameters from baseline timepoint (T0) to early-therapy T2 are prognostic of higher progression-free survival (PFS) rate at 6 months (PFS-6) from enrollment in patients treated with weekly or every-3-week paclitaxel regimens, who are receiving carboplatin with or without bevacizumab.***

IMAGING SECONDARY OBJECTIVES:

I. To determine whether larger changes in tumor perfusion parameters from baseline T0 to intermediate T1 and from T1 to T2 are prognostic of higher PFS-6 in patients treated with weekly or every-3-week paclitaxel regimens, who are receiving carboplatin with or without bevacizumab.*** II. To determine whether larger changes in tumor perfusion parameters values from T0 to T1, T0 to T2, and T1 to T2 are prognostic of better overall survival in all treatment arms.*** III. To assess the association between changes in tumor perfusion parameters before and after chemotherapy initiation (T0 to T1) and subsequent best tumor response according to standard anatomic Response Evaluation Criteria in Solid Tumors (RECIST).*** IV. To assess the association between tumor perfusion parameters before chemotherapy and subsequent best tumor response according to RECIST, PFS-6, and overall survival.*** V. To test the assumption that tumor perfusion parameters are reliable, user-independent, and reproducible parameters of tumor microvascular characteristics; a subgroup of 15 patients will have repeat computed tomography (CT) perfusion studies at the intermediate T1 time point.***

NOTE: ***Patients enrolled after February 8, 2012 must participate in the ACRIN 6695 component at ACRIN-qualified institutions.

OUTLINE: Patients are randomized to 1 of 2 treatment arms (beginning on 04-30-2012, the trial is no longer randomized and the chemotherapy regimen is selected and declared prior to enrolling in the study).

ARM I (adjuvant chemotherapy suboptimally debulked): Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses.

ARM II (neoadjuvant chemotherapy with interval cytoreductive surgery): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses. Patients undergo interval cytoreductive surgery between courses 3 and 4.

Patients in both arms may receive optional** bevacizumab IV over 30-90 minutes on day 1 beginning in course 2. Courses of bevacizumab repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients in Arm II receive bevacizumab during courses 2, 5, and 6 only.

NOTE: **Before enrolling onto this study, each patient chooses whether the study treatment will include concurrent and maintenance bevacizumab.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Primary Surgery and Neoadjuvant Chemotherapy with Interval Cytoreductive Surgery Patients:
* Patients must have measurable disease; at least one target lesion must have a minimum length of 1 cm in both the long and short axis (determined at the local site); for primary surgery patients, if no radiographic evidence of measurable disease is obtained prior to registration this can be based on surgical findings; imaging then would need to be completed in the 14 days between Gynecology Oncology Group (GOG) registration and chemotherapy initiation

  * After GOG registration, the American College of Radiology [ACR] Imaging Core Laboratory will confirm target lesion as required per protocol; the GOG-eligibility (RECIST) scan and baseline T0 perfusion CT scans will be reviewed prior to the intermediate T1 perfusion CT time point
* Primary Surgery Patients:
* Patients with a histologic diagnosis of epithelial ovarian cancer, peritoneal primary carcinoma or fallopian tube cancer, stage II -IV suboptimally debulked (any residual disease > 1 cm); International Federation of Gynecology and Obstetrics (FIGO) stage is assessed following the completion of initial abdominal surgery, appropriate imaging studies and with appropriate tissue available for histologic evaluation; the minimum surgery required is an abdominal surgery providing tissue for histologic evaluation and establishing and documenting the primary site and stage; if additional surgery was performed, it should have been in accordance with appropriate surgery for ovarian or peritoneal carcinoma described in the GOG Surgical Procedures Manual
* Neoadjuvant Chemotherapy (NAC) with Interval Cytoreductive Surgery (ICS) Patients:
* For patients undergoing NAC-ICS, a core tissue (not fine needle aspiration) biopsy is required; the tissue must be consistent with a Müllerian origin; patients will require documentation of at least stage II or extraovarian sites of disease acquired via imaging or surgery (without attempt at cytoreduction)
* Patients with the following histologic epithelial cell types are eligible: serous, endometrioid, clear cell, mucinous adenocarcinoma, undifferentiated carcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S.); however, the histologic features of the tumor must be compatible with a primary Müllerian epithelial adenocarcinoma; patients may have co-existing fallopian tube carcinoma in-situ so long as the primary origin of invasive tumor is ovarian, peritoneal or fallopian tube; of note, patients with clear cell and mucinous tumors will be eligible unless there is a higher priority protocol
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl; this ANC cannot have been induced or supported by granulocyte colony stimulating factors
* Platelets greater than or equal to 100,000/mcl
* Creatinine =< 1.5 x institutional upper limit normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Neuropathy (sensory or motor) less than or equal to Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Patients must have a GOG performance status of 0, 1, or 2
* Patients must be entered within 12 weeks of diagnostic/staging surgery
* Patients who have met the pre-entry requirements
* An approved informed consent and authorization permitting release of personal health information and must be signed by the patient or guardian
* Only applies for patients who elect to receive bevacizumab:

  * Patients in this trial may receive ovarian estrogen +/- progestin replacement therapy as indicated at the lowest effective dose(s) for control of menopausal symptoms at any time, but not high-dose progestins for management of anorexia while on protocol-directed therapy or prior to disease progression due to thrombophlebitis risk
  * Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thromboembolus) and a partial prothrombin time (PTT) < 1.2 times the upper limit of normal; (heparin, lovenox or alternative anticoagulants are acceptable)
  * All patients enrolled into GOG-0262 at sites where ACRIN 6695 is open will be enrolled in the advanced imaging protocol; patients receiving adjuvant or neoadjuvant chemotherapy are eligible for ACRIN 6695; the following sentence does not apply to those patients entered after 02/08/2012: if a patient declines to participate in the perfusion imaging portion of the protocol, a clinical rationale for declination of imaging form will be completed as part of the data submission for ACRIN 6695
* ACRIN 6695 Eligible Patients:

  * Confirmation of ACRIN 6695 eligibility after the baseline T0 perfusion computed tomography (CT) will be assessed by the ACR Imaging Core Lab: At least one target lesion must have a minimum length of 1 cm in both the long and short axis (as determined by the local site), at least half of the target lesion must have attenuation greater than or equal to 10 Hounsfield Units (HU) on the unenhanced CT, and at least half of the lesion must have maximum enhancement greater than or equal to 5 HU in the perfusion CT scan (as determined by the ACR Imaging Core Lab)

Exclusion Criteria:

* Patients with a current diagnosis of borderline epithelial ovarian tumor (formerly "tumors of low malignant potential") or recurrent invasive epithelial ovarian, primary peritoneal or fallopian tube cancer treated with surgery only (such as patients with stage I-A or I-B low grade epithelial ovarian or fallopian tube cancers) are not eligible; patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated, new invasive epithelial ovarian, peritoneal primary or fallopian tube cancer are eligible, provided that they have not received prior chemotherapy for any ovarian tumor
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor including neo-adjuvant chemotherapy for their ovarian, primary peritoneal or fallopian tube cancer; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients who have received any targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their epithelial ovarian, fallopian tube or peritoneal primary cancer
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, unless all of the following conditions are met: stage not greater than I-A, grade 1 or 2, no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO grade 3 lesions
* With the exception of non-melanoma skin cancer, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last five years or whose previous cancer treatment contraindicates this protocol therapy
* Patients with acute hepatitis or active infection that requires parenteral antibiotics
* Patients with clinically significant cardiovascular disease; this includes:

  * Myocardial infarction or unstable angina < 6 months prior to registration
  * New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Serious cardiac arrhythmia requiring medication; this does not include asymptomatic, atrial fibrillation with controlled ventricular rate
* Patients who are pregnant or nursing; patients of childbearing potential must agree to use contraceptive measures during study therapy and for at least six months after completion of bevacizumab therapy
* Patients who have received prior therapy with any anti-vascular endothelial growth factor (VEGF) drug, including bevacizumab
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study; the investigator should feel free to consult the Statistical and Data Center (SDC) randomization desk for uncertainty in this regard
* Patients with known allergy to cremophor or polysorbate 80
* Only applies to patients who elect to receive bevacizumab:
* Patients with serious non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days; patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study

  * Patients with CTCAE grade 2 or greater peripheral vascular disease (at least brief [< 24 hours] episodes of ischemia managed non-surgically and without permanent deficit)
  * Patients with a history of CVA within six months
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients with clinically significant proteinuria; urine protein should be screened by urine protein-creatinine ratio (UPCR); the UPCR has been found to correlate directly with the amount of protein excreted in a 24 hour urine collection; specifically, a UPCR of 1.0 is equivalent to 1.0 gram of protein in a 24-hour urine collection; obtain at least 4 ml of a random urine sample in a sterile container (does not have to be a 24-hour urine); send sample to lab with request for urine protein and creatinine levels (separate requests); the lab will measure protein concentration (mg/dL) and creatinine concentration (mg/dL); the UPCR is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL); patients must have a UPCR < 1.0 to allow participation in the study
* Patients with or with anticipation of invasive procedures as defined below:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of bevacizumab therapy (cycle 2)
  * Major surgical procedure anticipated during the course of the study; this includes, but is not limited to abdominal surgery (laparotomy or laparoscopy) prior to disease progression such as colostomy or enterostomy reversal, secondary cytoreductive surgery, or second look surgery; please consult with the SDC Randomization Desk prior to patient entry for any questions related to the classification of surgical procedures
  * Any tissue biopsy, such as a core biopsy, within 7 days prior to the first date of bevacizumab therapy (cycle 2)
* Patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration and/or nutrition
* Patients with metastasis tumor in the parenchyma of the liver or lungs with proximity to large vessels which could make the patients at high risk of lethal hemorrhage during treatment with bevacizumab (ie. hemoptysis, liver rupture)
* ACRIN 6695 Ineligible Patients:

  * Patients with contraindication to iodinated contrast for perfusion CT imaging
  * Patients who receive Metformin within 48 hours before perfusion CT imaging

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2026-07-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John K Chan, Principal Investigator — NRG Oncology
Locations (564):
- United States (559):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - John Muir Medical Center-Concord, Concord, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - GenesisCare USA - FGO, Fort Myers, Florida
  - Southeast Gynecologic Oncology Associates, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - The Watson Clinic, Lakeland, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Freeman Health System, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Luke's Hospital-Warren Campus, Phillipsburg, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Queens Hospital Center, Jamaica, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- South Korea (4):
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yongdong Severence Hospital, Seoul

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Chan JK, Brady MF, Penson RT, Huang H, Birrer MJ, Walker JL, DiSilvestro PA, Rubin SC, Martin LP, Davidson SA, Huh WK, O'Malley DM, Boente MP, Michael H, Monk BJ. Weekly vs. Every-3-Week Paclitaxel and Carboplatin for Ovarian Cancer. N Engl J Med. 2016 Feb 25;374(8):738-48. doi: 10.1056/NEJMoa1505067. PMID 26933849
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Newly diagnosed women with high-risk early stage or advanced stage epithelial ovarian cancer enrolled from September 27, 2010 to February 8, 2012.These women were randomly assigned to receive either carboplatin (AUC 6) combined with either paclitaxel 175 mg/m2 q 21 days or paclitaxel 80mg/m2 on days 1, 8 and 15. Bevacizumab was optional.
Pre-assignment Details: 112 additional women, whose treatment was not randomized, enrolled onto this study in order to evaluate whether findings from perfusion imaging are prognostic. This report focuses on the randomized treatment component of this study.
Period: Overall Study
Arm/Group | Arm I (Adjuvant Chemotherapy Suboptimally Debulked) | Arm II (Neoadjuvant Chemotherapy)
Started | 346 | 346
Completed | 346 | 346
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Newly diagnosed women with high-risk early stage or advanced stage epithelial ovarian cancer.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Adjuvant Chemotherapy Suboptimally Debulked) | Arm II (Neoadjuvant Chemotherapy) | Total
Number analyzed (Participants) | 346 | 346 | 692
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 214 | 217 | 431
  >=65 years | 132 | 129 | 261
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 346 | 346 | 692
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 0 | 1
  United States | 345 | 345 | 690
  South Korea | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: First progression or death for weekly paclitaxel treatment relative to standard 3 week paclitaxel. Progression is defined using response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: The timeframe is from enrollment onto the study up to 3 years following enrollment.
Population: Whole sample
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Adjuvant Chemotherapy Suboptimally Debulked) | Arm II (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 346 | 346
months | 14.7 [13.5 to 15.8] | 14.0 [12.7 to 15.2]
Statistical Analysis 1: Comparison: Arm I (Adjuvant Chemotherapy Suboptimally Debulked) vs Arm II (Neoadjuvant Chemotherapy); Estimated hazard of first progression or death for weekly paclitaxel treatment relative to standard 3 week paclitaxel; Test type: Superiority; Hazard Ratio (HR) = .89, 95% CI 2-sided [.74 to 1.06]

2. Secondary Outcome: Median Duration of First Quartile Survival
Description: First Quartile Overall Survival
Time Frame: The timeframe is from enrollment onto the study up to 3 years after enrollment
Population: Whole sample
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Adjuvant Chemotherapy Suboptimally Debulked) | Arm II (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 346 | 346
months | 23.2 [20.1 to 26.3] | 24 [19.8 to 26.0]
Statistical Analysis 1: Comparison: Arm I (Adjuvant Chemotherapy Suboptimally Debulked) vs Arm II (Neoadjuvant Chemotherapy); Test type: Superiority; Hazard Ratio (HR) = .94, 95% CI 2-sided [.72 to 1.23]

3. Secondary Outcome: Quality of Life Score as Measured by Functional Assessment of Cancer Therapy-Ovary-Total Outcome Index (Fact-O TOI)
Description: Mean quality of life score after 6 cycles of study treatment estimated from a mixed model. The FACT-O-TOI is composed of three subscales: Physical Well Being (PWB) (7 Items), Functional Well Being (FWB) (7 items), and Ovarian Cancer Subscale (OCS) (12 items). Each item in the FACT-O TOI are scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). A subscale score is computed as long as more than 50% of subscale items have been answered. A Total score of the FACT-O TOI is the summation of the three subscale scores; if more than 80% of the FACT-O TOI items provide valid responses and all three subscales have valid scores. A score of the FACT-O TOI is ranged 0-104 with a larger score indicating a more preferred state of health-related quality of life (HRQOL)
Time Frame: 18 weeks after enrolling on the study, which is the time it takes to complete 6 cycles of treatment plus 3 weeks
Population: All individuals who did not opt for neo-adjuvant treatment and completed a baseline FACT-O TOI assessment and at least one follow-up assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Arm I (Adjuvant Chemotherapy Suboptimally Debulked) | Arm II (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 292 | 287
Units on a Scale | 70.9 (1.42) | 68.2 (1.59)

4. Other Pre Specified Outcome: Changes in the Tumor Perfusion Parameters as Quantified by Vascularity or Blood Volume; Perfusion or Blood Flow; Mean Transit Time; and Microvascular Permeability or Permeability Surface Area Product
Time Frame: Baseline (T0) up to 10 days after the start of course 2 (T2)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs were assessed from the date of treatment initiation up to 30 days after the last cycle of treatment.
Arm/Group | Arm I (Adjuvant Chemotherapy Suboptimally Debulked) | Arm II (Neoadjuvant Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 122/346 | 167/346
Other Adverse Events (participants affected / at risk) | 343/346 | 340/346
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Adjuvant Chemotherapy Suboptimally Debulked) (N=346) | Arm II (Neoadjuvant Chemotherapy) (N=346)
Hemolytic Uremic Syndrome (Blood and lymphatic system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 10 | 8
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 2 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 0 | 1
Dry Eye (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 1 | 0
Colonic Obstruction (Gastrointestinal disorders) | 1 | 1
Colonic Perforation (Gastrointestinal disorders) | 0 | 2
Colonic Fistula (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 5
Duodenal Perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 7
Small Intestinal Obstruction (Gastrointestinal disorders) | 8 | 13
Abdominal Pain (Gastrointestinal disorders) | 6 | 7
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Obstruction Gastric (Gastrointestinal disorders) | 1 | 2
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 2
Ileal Perforation (Gastrointestinal disorders) | 1 | 1
Ileal Obstruction (Gastrointestinal disorders) | 1 | 0
Ileal Fistula (Gastrointestinal disorders) | 1 | 0
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Fistula (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Rectal Pain (Gastrointestinal disorders) | 1 | 0
Gastric Perforation (Gastrointestinal disorders) | 0 | 1
Gastric Fistula (Gastrointestinal disorders) | 0 | 1
Esophageal Ulcer (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Jejunal Obstruction (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Multi-Organ Failure (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Death Nos (General disorders) | 1 | 1
Fever (General disorders) | 1 | 3
Infusion Related Reaction (General disorders) | 0 | 2
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0
Infections And Infestations - Other (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 1
Splenic Infection (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 5
Pleural Infection (Infections and infestations) | 1 | 0
Pelvic Infection (Infections and infestations) | 1 | 3
Lung Infection (Infections and infestations) | 0 | 2
Kidney Infection (Infections and infestations) | 0 | 1
Endocarditis Infective (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 2
Catheter Related Infection (Infections and infestations) | 0 | 5
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Bladder Infection (Infections and infestations) | 0 | 1
Anorectal Infection (Infections and infestations) | 0 | 1
Abdominal Infection (Infections and infestations) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 4
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Stomal Ulcer (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Wound Complication (Injury, poisoning and procedural complications) | 2 | 0
Platelet Count Decreased (Investigations) | 0 | 2
Neutrophil Count Decreased (Investigations) | 7 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient Ischemic Attacks (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 2
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Urinary Fistula (Renal and urinary disorders) | 0 | 1
Renal Calculi (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal Fistula (Reproductive system and breast disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 2 | 1
Thromboembolic Event (Vascular disorders) | 1 | 9
Peripheral Ischemia (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 5 | 0
Hematoma (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Adjuvant Chemotherapy Suboptimally Debulked) (N=346) | Arm II (Neoadjuvant Chemotherapy) (N=346)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 3 | 2
Lymph Node Pain (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 8 | 13
Anemia (Blood and lymphatic system disorders) | 324 | 336
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Bone Marrow Hypocellular (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 6
Atrial Fibrillation (Cardiac disorders) | 0 | 6
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 3
Sinus Bradycardia (Cardiac disorders) | 1 | 2
Palpitations (Cardiac disorders) | 10 | 24
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Disorders - Other (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 1
Ventricular Arrhythmia (Cardiac disorders) | 0 | 2
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 2 | 0
Sinus Tachycardia (Cardiac disorders) | 12 | 17
Chest Pain - Cardiac (Cardiac disorders) | 5 | 6
Middle Ear Inflammation (Ear and labyrinth disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 6 | 10
Tinnitus (Ear and labyrinth disorders) | 28 | 20
Hearing Impaired (Ear and labyrinth disorders) | 14 | 13
Ear Pain (Ear and labyrinth disorders) | 8 | 10
External Ear Inflammation (Ear and labyrinth disorders) | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 3
Hyperthyroidism (Endocrine disorders) | 1 | 1
Endocrine Disorders - Other (Endocrine disorders) | 2 | 1
Cushingoid (Endocrine disorders) | 0 | 1
Eye Disorders - Other (Eye disorders) | 10 | 10
Watering Eyes (Eye disorders) | 11 | 15
Flashing Lights (Eye disorders) | 3 | 3
Eye Pain (Eye disorders) | 4 | 1
Glaucoma (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 2
Photophobia (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 2
Retinal Vascular Disorder (Eye disorders) | 1 | 0
Blurred Vision (Eye disorders) | 47 | 51
Dry Eye (Eye disorders) | 3 | 9
Floaters (Eye disorders) | 12 | 11
Vitreous Hemorrhage (Eye disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 11 | 14
Dyspepsia (Gastrointestinal disorders) | 21 | 28
Dry Mouth (Gastrointestinal disorders) | 12 | 10
Colonic Obstruction (Gastrointestinal disorders) | 2 | 0
Colonic Perforation (Gastrointestinal disorders) | 2 | 1
Colonic Fistula (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 6 | 2
Colonic Hemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 226 | 214
Diarrhea (Gastrointestinal disorders) | 146 | 153
Vomiting (Gastrointestinal disorders) | 133 | 115
Bloating (Gastrointestinal disorders) | 32 | 21
Stomach Pain (Gastrointestinal disorders) | 7 | 3
Salivary Duct Inflammation (Gastrointestinal disorders) | 0 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Anal Hemorrhage (Gastrointestinal disorders) | 3 | 1
Rectal Ulcer (Gastrointestinal disorders) | 0 | 1
Anal Mucositis (Gastrointestinal disorders) | 1 | 0
Rectal Fistula (Gastrointestinal disorders) | 0 | 3
Rectal Mucositis (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 139 | 138
Proctitis (Gastrointestinal disorders) | 0 | 1
Periodontal Disease (Gastrointestinal disorders) | 3 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 16 | 7
Oral Dysesthesia (Gastrointestinal disorders) | 3 | 3
Mucositis Oral (Gastrointestinal disorders) | 76 | 93
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 14 | 16
Anal Pain (Gastrointestinal disorders) | 0 | 4
Oral Hemorrhage (Gastrointestinal disorders) | 15 | 8
Ileus (Gastrointestinal disorders) | 5 | 5
Ileal Fistula (Gastrointestinal disorders) | 1 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 5 | 7
Gastric Hemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 7 | 3
Oral Pain (Gastrointestinal disorders) | 14 | 16
Abdominal Distension (Gastrointestinal disorders) | 25 | 15
Nausea (Gastrointestinal disorders) | 239 | 215
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Gastroparesis (Gastrointestinal disorders) | 2 | 3
Gastrointestinal Fistula (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 21 | 27
Rectal Pain (Gastrointestinal disorders) | 1 | 8
Lip Pain (Gastrointestinal disorders) | 1 | 0
Gastric Fistula (Gastrointestinal disorders) | 0 | 1
Esophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 2 | 1
Fecal Incontinence (Gastrointestinal disorders) | 0 | 3
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 8 | 10
Hemorrhoids (Gastrointestinal disorders) | 14 | 20
Ascites (Gastrointestinal disorders) | 14 | 4
Toothache (Gastrointestinal disorders) | 11 | 1
Jejunal Obstruction (Gastrointestinal disorders) | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 1 | 0
Esophageal Pain (Gastrointestinal disorders) | 0 | 2
Dental Caries (Gastrointestinal disorders) | 4 | 2
Flatulence (Gastrointestinal disorders) | 11 | 10
Gastritis (Gastrointestinal disorders) | 5 | 5
General Disorders And Administration Site Conditio (General disorders) | 3 | 8
Pain (General disorders) | 93 | 86
Neck Edema (General disorders) | 1 | 1
Malaise (General disorders) | 8 | 6
Localized Edema (General disorders) | 5 | 4
Irritability (General disorders) | 1 | 0
Injection Site Reaction (General disorders) | 0 | 2
Infusion Site Extravasation (General disorders) | 0 | 2
Flu Like Symptoms (General disorders) | 13 | 8
Edema Trunk (General disorders) | 2 | 3
Non-Cardiac Chest Pain (General disorders) | 14 | 11
Edema Limbs (General disorders) | 54 | 65
Facial Pain (General disorders) | 4 | 4
Edema Face (General disorders) | 4 | 3
Fatigue (General disorders) | 293 | 300
Fever (General disorders) | 26 | 38
Gait Disturbance (General disorders) | 5 | 9
Chills (General disorders) | 14 | 23
Infusion Related Reaction (General disorders) | 12 | 15
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 1 | 0
Hepatic Pain (Hepatobiliary disorders) | 1 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 18 | 11
Cytokine Release Syndrome (Immune system disorders) | 1 | 0
Immune System Disorders - Other (Immune system disorders) | 1 | 1
Infections And Infestations - Other (Infections and infestations) | 12 | 11
Wound Infection (Infections and infestations) | 9 | 6
Upper Respiratory Infection (Infections and infestations) | 19 | 16
Tooth Infection (Infections and infestations) | 8 | 9
Stoma Site Infection (Infections and infestations) | 0 | 1
Vulval Infection (Infections and infestations) | 3 | 2
Skin Infection (Infections and infestations) | 5 | 17
Sinusitis (Infections and infestations) | 15 | 16
Sepsis (Infections and infestations) | 1 | 3
Salivary Gland Infection (Infections and infestations) | 0 | 1
Rhinitis Infective (Infections and infestations) | 4 | 1
Rash Pustular (Infections and infestations) | 1 | 0
Pleural Infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2
Peritoneal Infection (Infections and infestations) | 0 | 1
Peripheral Nerve Infection (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Papulopustular Rash (Infections and infestations) | 3 | 3
Otitis Externa (Infections and infestations) | 1 | 1
Nail Infection (Infections and infestations) | 4 | 7
Mucosal Infection (Infections and infestations) | 4 | 4
Pelvic Infection (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 3 | 3
Laryngitis (Infections and infestations) | 1 | 3
Kidney Infection (Infections and infestations) | 1 | 0
Hepatitis Viral (Infections and infestations) | 1 | 0
Eye Infection (Infections and infestations) | 0 | 2
Esophageal Infection (Infections and infestations) | 1 | 0
Duodenal Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 2
Conjunctivitis Infective (Infections and infestations) | 0 | 1
Gum Infection (Infections and infestations) | 2 | 1
Vaginal Infection (Infections and infestations) | 9 | 5
Urinary Tract Infection (Infections and infestations) | 44 | 52
Catheter Related Infection (Infections and infestations) | 1 | 5
Bronchial Infection (Infections and infestations) | 5 | 3
Enterocolitis Infectious (Infections and infestations) | 4 | 3
Bladder Infection (Infections and infestations) | 3 | 8
Lip Infection (Infections and infestations) | 1 | 0
Anorectal Infection (Infections and infestations) | 1 | 1
Abdominal Infection (Infections and infestations) | 1 | 3
Injury, Poisoning And Procedural Complications - O (Injury, poisoning and procedural complications) | 2 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 3 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 5 | 7
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 | 4
Vaginal Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 2
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 2 | 3
Tracheal Obstruction (Injury, poisoning and procedural complications) | 0 | 1
Intestinal Stoma Site Bleeding (Injury, poisoning and procedural complications) | 0 | 1
Stomal Ulcer (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 8 | 9
Wound Complication (Injury, poisoning and procedural complications) | 17 | 13
Intraoperative Musculoskeletal Injury (Injury, poisoning and procedural complications) | 1 | 0
Burn (Injury, poisoning and procedural complications) | 2 | 2
Bruising (Injury, poisoning and procedural complications) | 20 | 17
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Investigations - Other (Investigations) | 15 | 14
Weight Loss (Investigations) | 56 | 48
Weight Gain (Investigations) | 53 | 39
Serum Amylase Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 257 | 274
Pancreatic Enzymes Decreased (Investigations) | 0 | 2
Lymphocyte Count Decreased (Investigations) | 18 | 36
Lipase Increased (Investigations) | 1 | 0
Inr Increased (Investigations) | 5 | 9
Hemoglobin Increased (Investigations) | 1 | 1
Ggt Increased (Investigations) | 2 | 5
Ejection Fraction Decreased (Investigations) | 1 | 0
Creatinine Increased (Investigations) | 24 | 34
Cholesterol High (Investigations) | 6 | 5
Neutrophil Count Decreased (Investigations) | 325 | 331
Urine Output Decreased (Investigations) | 0 | 1
Cardiac Troponin I Increased (Investigations) | 1 | 0
Cpk Increased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 7 | 8
White Blood Cell Decreased (Investigations) | 321 | 332
Aspartate Aminotransferase Increased (Investigations) | 40 | 42
Alkaline Phosphatase Increased (Investigations) | 41 | 47
Alanine Aminotransferase Increased (Investigations) | 38 | 39
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 6
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 11 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 10 | 22
Hyponatremia (Metabolism and nutrition disorders) | 57 | 63
Hypomagnesemia (Metabolism and nutrition disorders) | 68 | 86
Hypokalemia (Metabolism and nutrition disorders) | 60 | 66
Hypoglycemia (Metabolism and nutrition disorders) | 14 | 15
Hypocalcemia (Metabolism and nutrition disorders) | 28 | 48
Hypoalbuminemia (Metabolism and nutrition disorders) | 49 | 65
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 4
Hypernatremia (Metabolism and nutrition disorders) | 9 | 10
Hypermagnesemia (Metabolism and nutrition disorders) | 4 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 16 | 15
Hyperglycemia (Metabolism and nutrition disorders) | 73 | 82
Hypercalcemia (Metabolism and nutrition disorders) | 17 | 13
Glucose Intolerance (Metabolism and nutrition disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 36 | 38
Anorexia (Metabolism and nutrition disorders) | 102 | 116
Acidosis (Metabolism and nutrition disorders) | 2 | 0
Superficial Soft Tissue Fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 80 | 69
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 21 | 15
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 91 | 75
Musculoskeletal Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscle Weakness Trunk (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 15 | 13
Muscle Weakness Right-Sided (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint Range Of Motion Decreased Cervical Spine (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 4 | 7
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 3
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 35 | 44
Flank Pain (Musculoskeletal and connective tissue disorders) | 10 | 3
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 7 | 14
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 33 | 25
Back Pain (Musculoskeletal and connective tissue disorders) | 70 | 54
Arthritis (Musculoskeletal and connective tissue disorders) | 19 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 119 | 83
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 4 | 8
Neoplasms Benign, Malignant And Unspecified (Including cysts and polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Nervous System Disorders - Other (Nervous system disorders) | 3 | 6
Tremor (Nervous system disorders) | 4 | 9
Transient Ischemic Attacks (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 244 | 233
Peripheral Motor Neuropathy (Nervous system disorders) | 19 | 20
Paresthesia (Nervous system disorders) | 19 | 24
Nystagmus (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 5 | 6
Memory Impairment (Nervous system disorders) | 20 | 20
Lethargy (Nervous system disorders) | 0 | 1
Movements Involuntary (Nervous system disorders) | 5 | 3
Hypersomnia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 116 | 112
Facial Nerve Disorder (Nervous system disorders) | 0 | 1
Extrapyramidal Disorder (Nervous system disorders) | 2 | 0
Radiculitis (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 42 | 58
Sinus Pain (Nervous system disorders) | 5 | 6
Dysesthesia (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 8 | 6
Dizziness (Nervous system disorders) | 61 | 66
Concentration Impairment (Nervous system disorders) | 1 | 4
Cognitive Disturbance (Nervous system disorders) | 7 | 5
Ataxia (Nervous system disorders) | 3 | 4
Amnesia (Nervous system disorders) | 1 | 1
Akathisia (Nervous system disorders) | 1 | 1
Psychiatric Disorders - Other (Psychiatric disorders) | 2 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 8 | 6
Libido Decreased (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 90 | 85
Depression (Psychiatric disorders) | 66 | 66
Delirium (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 5 | 5
Anxiety (Psychiatric disorders) | 60 | 68
Agitation (Psychiatric disorders) | 4 | 7
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 4 | 12
Urine Discoloration (Renal and urinary disorders) | 0 | 1
Urinary Urgency (Renal and urinary disorders) | 9 | 11
Urinary Tract Obstruction (Renal and urinary disorders) | 2 | 3
Urinary Retention (Renal and urinary disorders) | 4 | 7
Urinary Incontinence (Renal and urinary disorders) | 13 | 17
Urinary Tract Pain (Renal and urinary disorders) | 16 | 18
Urinary Frequency (Renal and urinary disorders) | 14 | 34
Urinary Fistula (Renal and urinary disorders) | 0 | 1
Renal Calculi (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 47 | 55
Hematuria (Renal and urinary disorders) | 11 | 13
Cystitis Noninfective (Renal and urinary disorders) | 0 | 3
Chronic Kidney Disease (Renal and urinary disorders) | 2 | 6
Bladder Spasm (Renal and urinary disorders) | 3 | 2
Acute Kidney Injury (Renal and urinary disorders) | 3 | 2
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 3 | 2
Vaginal Pain (Reproductive system and breast disorders) | 4 | 7
Vaginal Hemorrhage (Reproductive system and breast disorders) | 4 | 7
Vaginal Fistula (Reproductive system and breast disorders) | 1 | 4
Vaginal Dryness (Reproductive system and breast disorders) | 8 | 6
Perineal Pain (Reproductive system and breast disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 11 | 8
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 7 | 17
Vaginal Inflammation (Reproductive system and breast disorders) | 1 | 3
Genital Edema (Reproductive system and breast disorders) | 0 | 2
Dyspareunia (Reproductive system and breast disorders) | 5 | 4
Breast Pain (Reproductive system and breast disorders) | 1 | 3
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 15 | 15
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 27 | 25
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 22 | 24
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pharyngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 42 | 45
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 20 | 25
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 89 | 131
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 120 | 131
Cough (Respiratory, thoracic and mediastinal disorders) | 76 | 90
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 39 | 46
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 28 | 33
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2
Skin Ulceration (Skin and subcutaneous tissue disorders) | 10 | 4
Skin Induration (Skin and subcutaneous tissue disorders) | 2 | 3
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 | 9
Scalp Pain (Skin and subcutaneous tissue disorders) | 5 | 2
Rash Acneiform (Skin and subcutaneous tissue disorders) | 18 | 24
Purpura (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 22
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 1
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 5
Pain Of Skin (Skin and subcutaneous tissue disorders) | 3 | 7
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 43 | 74
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Nail Ridging (Skin and subcutaneous tissue disorders) | 12 | 9
Nail Loss (Skin and subcutaneous tissue disorders) | 6 | 20
Nail Discoloration (Skin and subcutaneous tissue disorders) | 13 | 33
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 5 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 24 | 36
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Body Odor (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 258 | 235
Social Circumstances - Other (Social circumstances) | 6 | 2
Menopause (Social circumstances) | 1 | 0
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 8 | 11
Vascular Disorders - Other (Vascular disorders) | 1 | 4
Thromboembolic Event (Vascular disorders) | 23 | 21
Superficial Thrombophlebitis (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1
Peripheral Ischemia (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 2 | 2
Lymphedema (Vascular disorders) | 8 | 12
Hypotension (Vascular disorders) | 13 | 14
Hypertension (Vascular disorders) | 136 | 122
Hot Flashes (Vascular disorders) | 44 | 39
Hematoma (Vascular disorders) | 4 | 3
Flushing (Vascular disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less